CLINICAL TRIAL: NCT00307437
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial Evaluating the Efficacy and Safety of CNTO 1275 in the Treatment of Subjects With Moderate to Severe Plaque-type Psoriasis.
Brief Title: A Study of the Safety and Efficacy of Ustekinumab (CNTO 1275) in Patients With Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor Research & Development, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR006325; C0743T09 (Other: Centocor R&D, USA); 2005-003530-17 (EudraCT Number)
Record Dates: First submitted 2006-03-24; First posted 2006-03-28 (Estimated); Results first posted 2012-11-02 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Psoriasis
Keywords: Moderate to Severe Plaque-Type Psoriasis; interleukin 23; IL-12; interleukin-12; interleukin-23; CNTO1275; biologic; Psoriasis; CNTO 1275; IL23; interleukin 12; IL-23; IL12; ustekinumab
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Ustekinumab (CNTO 1275) 45 or 90 mg
- Group II: Ustekinumab 45 mg (Experimental)
  Interventions: Drug: Ustekinumab (CNTO 1275) 45 mg
- Group III: Ustekinumab 90 mg (Experimental)
  Interventions: Drug: Ustekinumab (CNTO 1275) 90 mg

INTERVENTIONS:
Drug: Placebo; Ustekinumab (CNTO 1275) 45 or 90 mg — Placebo at Weeks 0 and 4 and blinded SC injections of ustekinumab, 45 or 90 mg, at Weeks 12 and 16; followed by a dosing regimen to be determined by patient's response status for Weeks 28 to 52; followed by unblinded dosing that may be adjusted at the investigator's discretion for Weeks 52 to 264
  Arms: Group I: Placebo
Drug: Ustekinumab (CNTO 1275) 45 mg — Ustekinumab, 45 mg, at Weeks 0 and 4 and every 12 weeks for Weeks 16 to 28. Followed by a dosing regimen to be determined by patient's response status for Weeks 28 to 52; followed by unblinded dosing that may be adjusted at the investigator's discretion for Weeks 52 to 264
  Arms: Group II: Ustekinumab 45 mg
Drug: Ustekinumab (CNTO 1275) 90 mg — Ustekinumab, 90 mg, at Weeks 0 and 4 and every 12 weeks for Weeks 16 to 28. Followed by a dosing regimen to be determined by patient's response status for Weeks 28 to 52; followed by unblinded dosing that may be adjusted at the investigator's discretion for Weeks 52 to 264
  Arms: Group III: Ustekinumab 90 mg

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of ustekinumab (CNTO 1275) in the treatment of patients with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
Although numerous therapeutic options exist for the treatment of psoriasis, there is still a significant unmet medical need due to the limited effectiveness and/or significant side effect profile of current treatment options. Preclinical studies and early phase clinical studies suggest that interleukins-12 and -23, two molecules that are part of the communication network in the immune system, may play an important role in psoriasis. Ustekinumab (CNTO 1275) is a monoclonal antibody directed against interleukins -12 and -23. This is a randomized (study drug assigned by chance like flipping a coin), double blind (neither physician nor patient knows the name of the assigned drug), parallel-group, multicenter study to determine the effectiveness and safety of two different doses of ustekinumab (CNTO 1275) administered subcutaneously (under the skin) as compared with placebo in patients with moderate to severe plaque-type psoriasis (the most common type of psoriasis). The hypothesis is that ustekinumab (CNTO 1275) will be more effective in treatment of psoriasis than placebo, that the improvement in psoriasis will result in an improved quality of life for treated patients and that ustekinumab (CNTO 1275) will be generally well tolerated. Patients will receive ustekinumab (CNTO 1275), 45 or 90 mg, or placebo administered subcutaneously at weeks 0 and 4 weeks then every 12 weeks thereafter until week 52. For patients who partially respond to the starting regimen, the dosing interval may be adjusted to every 8 weeks. Patients will enter long term extension portion of the study at week 52 during which patients will continue to receive treatment with ustekinumab (CNTO 1275) and will be followed for a total of up to 264 weeks from the initial (week 0) administration of study agent.

The dose of ustekinumab (CNTO 1275) will be 45 or 90 mg or placebo administered subcutaneously at weeks 0 and 4 weeks then every 12 weeks thereafter. For patients who partially respond to the starting regimen, the dosing interval may be adjusted to every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Plaque-type psoriasis diagnosed >= 6 months prior
* Plaque-type psoriasis covering at least 10% of total body surface areas
* Psoriasis area-and-severity index score of >=12 at screening and baseline
* Considered by treating dermatologist to be a candidate for phototherapy or systemic treatment of psoriasis
* Women of childbearing potential and all men must agree to use adequate birth control measures throughout the trials and for 12 months following the last injection of study agent
* Have no history of latent or active tuberculosis (TB)

Exclusion Criteria:

* Currently have nonplaque forms of psoriasis or drug-induced psoriasis
* Women who are pregnant or nursing, or men and women planning pregnancy while enrolled in the study
* Patients who have used any therapeutic agent targeted at reducing IL-12 or IL-23
* Patients who have had a Bacillus Calmette-Guerin (BCG) vaccination within the previous 12 months prior to screening
* Patients who have a history of chronic or recurrent infectious disease or who have or have had a serious infection requiring hospitalization or intravenous antibiotics within the previous 2 months prior to screening
* Patients who have or ever have had a nontuberculous mycobacterial infection or opportunistic infection
* Patients known to be infected with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Patients who have current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease
* Patients with a malignancy or who have a history of malignancy (with the exception of certain skin cancers and pre-invasive cervical cancer)
* Patients participating in another trial using an investigational agent or procedure
* Systemic immunosuppressants within 4 weeks of the first administration of study agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1230 (Actual)
Dates: Start 2005-05; Primary Completion 2006-12 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (62):
- United States (28):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - La Jolla, California
  - Los Angeles, California
  - San Diego, California
  - Jacksonville, Florida
  - Miami, Florida
  - Normal, Illinois
  - Skokie, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Andover, Massachusetts
  - Boston, Massachusetts
  - Port Huron, Michigan
  - St Louis, Missouri
  - Las Vegas, Nevada
  - New Brunswick, New Jersey
  - New York, New York
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Plymouth Meeting, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
- Austria (3):
  - Graz
  - Innsbruck
  - Vienna
- Canada (16):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Moncton, New Brunswick
  - Halifax, Nova Scotia
  - Barrie, Ontario
  - Hamilton, Ontario
  - London, Ontario
  - North Bay, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec
  - Sherbrooke, Quebec
- Nice, France
- Germany (9):
  - Berlin
  - Brandenburg
  - Dresden
  - Erlangen
  - Frankfurt
  - Hamburg
  - Kiel
  - Mainz
  - München
- Switzerland (2):
  - Geneva
  - Zurich
- United Kingdom (3):
  - London
  - Salford
  - Southampton Trials Carried Out

REFERENCES:
- [Derived] Ghosh S, Gensler LS, Yang Z, Gasink C, Chakravarty SD, Farahi K, Ramachandran P, Ott E, Strober BE. Ustekinumab Safety in Psoriasis, Psoriatic Arthritis, and Crohn's Disease: An Integrated Analysis of Phase II/III Clinical Development Programs. Drug Saf. 2019 Jun;42(6):751-768. doi: 10.1007/s40264-019-00797-3. PMID 30739254
- [Derived] Papp KA, Langley RG, Lebwohl M, Krueger GG, Szapary P, Yeilding N, Guzzo C, Hsu MC, Wang Y, Li S, Dooley LT, Reich K; PHOENIX 2 study investigators. Efficacy and safety of ustekinumab, a human interleukin-12/23 monoclonal antibody, in patients with psoriasis: 52-week results from a randomised, double-blind, placebo-controlled trial (PHOENIX 2). Lancet. 2008 May 17;371(9625):1675-84. doi: 10.1016/S0140-6736(08)60726-6. PMID 18486740

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this trial, 1230 participants were randomized to either placebo or ustekinumab (CNTO 1275). There were 70 sites in North America and Europe.
Pre-assignment Details: 2 participants from placebo group (in controlled period [CP]) after completing the CP did not crossover to the Placebo -> Ustekinumab 90 mg (after CP) treatment group and they are not included in this group (after CP). Thus, 1199 participants completed the 1st period (CP); however, only 1197 participants started the 2nd period (after CP).
Groups:
- Placebo (CP): Controlled period (Week 0-12) - Placebo group
- Ustekinumab 45 mg (CP): Controlled period (Week 0-12) - Ustekinumab 45 mg group
- Ustekinumab 90 mg (CP): Controlled period (Week 0-12) - Ustekinumab 90 mg group
- Placebo -> Ustekinumab 45 mg (After CP): After Controlled period (Week 12-264) - patients receiving Placebo at Weeks 0 and 4 -> receiving ustekinumab 45 mg q12wk or q8wk from Week 12 to Week 244. Some patients in this group dose escalated from ustekinumab 45 mg to 90 mg after Week 52.
- Placebo -> Ustekinumab 90 mg (After CP): After Controlled period (Week 12-264) - patients receiving Placebo at Weeks 0 and 4 -> receiving ustekinumab 90 mg q12wk or q8wk from Week 12 to Week 244.
- Ustekinumab 45 mg (After CP): After Controlled period (Week 12-264) - patients receiving ustekinumab 45 mg at Weeks 0 and 4 -> receiving ustekinumab 45 mg q12wk or q8wk from Week 16 to Week 244. Some patients in this group dose escalated from ustekinumab 45 mg to 90 mg after Week 52.
- Ustekinumab 90 mg (After CP): After Controlled period (Week 12-264) - patients receiving ustekinumab 90 mg at Weeks 0 and 4 -> receiving ustekinumab 90 mg q12wk or q8wk from Week 16 to Week 244.
Period: Controlled Period
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP) | Placebo -> Ustekinumab 45 mg (After CP) | Placebo -> Ustekinumab 90 mg (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Started | 410 | 409 | 411 | 0 ("0" in column indicates this reporting group is not relevant to Control Period.) | 0 ("0" in column indicates this reporting group is not relevant to Control Period.) | 0 ("0" in column indicates this reporting group is not relevant to Control Period.) | 0 ("0" in column indicates this reporting group is not relevant to Control Period.)
Completed | 394 | 403 | 402 | 0 | 0 | 0 | 0
Not Completed | 16 | 6 | 9 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 2 | 5 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 5 | 1 | 3 | 0 | 0 | 0 | 0
Period: After Controlled Period
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP) | Placebo -> Ustekinumab 45 mg (After CP) | Placebo -> Ustekinumab 90 mg (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Started | 0 ("0" in column indicates this reporting group is not relevant to after Control Period.) | 0 ("0" in column indicates this reporting group is not relevant to after Control Period.) | 0 ("0" in column indicates this reporting group is not relevant to after Control Period.) | 197 | 195 (2 participants from placebo group in CP did not crossover to this group after CP.) | 403 | 402
Completed | 0 | 0 | 0 | 139 | 140 | 281 | 289
Not Completed | 0 | 0 | 0 | 58 | 55 | 122 | 113
Not completed — Adverse Event | 0 | 0 | 0 | 18 | 16 | 31 | 40
Not completed — Death | 0 | 0 | 0 | 3 | 1 | 1 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 15 | 17 | 37 | 24
Not completed — Lost to Follow-up | 0 | 0 | 0 | 7 | 12 | 13 | 18
Not completed — Other | 0 | 0 | 0 | 15 | 9 | 40 | 28

BASELINE CHARACTERISTICS:
Groups:
- Group I: Placebo: Placebo participants received placebo at Weeks 0 and 4. At Weeks 12 and 16, placebo crossed over to receive ustekinumab 45 mg or 90 mg. Treatments after Week 16 were dependent on clinical response.
- Group II: Ustekinumab 45 mg: Participants received ustekinumab 45 mg at Weeks 0, 4 and 16. Treatments after Week 16 were dependent on clinical response. At Week 28, participants who achieved a greater than and equal to 50 percentage but less than 75 percentage improvement in PASI were re-randomized to continue 45 mg every 12 week or dose adjust to 45 mg every 8 week dosing.
- Group III: Ustekinumab 90 mg: Participants received ustekinumab 90 mg at Weeks 0, 4 and 16. Treatments after Week 16 were dependent on clinical response. At Week 28, participants who achieved a greater than and equal 50 percentage but less than 75 percentage improvement in PASI were re-randomized to continue 90 mg every 12 week or dose adjust to 90 mg every 8 week dosing.
- Total: Total of all reporting groups
Arm/Group | Group I: Placebo | Group II: Ustekinumab 45 mg | Group III: Ustekinumab 90 mg | Total
Number analyzed (Participants) | 410 | 409 | 411 | 1230
Age Continuous [Mean (Standard Deviation); unit: years] | 47.0 (12.47) | 45.1 (12.06) | 46.6 (12.14) | 46.2 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 126 | 137 | 390
  Male | 283 | 283 | 274 | 840

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Psoriasis Area and Severity Index (PASI) Score of 75 Percent or Above at Week 12
Description: Number of participants achieving greater than or equal to 75 percent improvement in PASI at Week 12. PASI is a widely used tool for the measurement of severity of psoriasis. This is a test of how bad a person's psoriasis is. The scale combines redness, scaling, and thickness, as well as overall body involvement to determine the PASI score. The scale ranges from 0 (best) to 72 (worst).
Time Frame: Week 0 to Week 12
Population: Intent to treat. All participants randomized were included in the analysis according to the assigned treatment groups. Participant is considered a non- responder if the participant has used any pre-specified prohibited medications or discontinued due to lack of efficacy or had missing data at Week 12.
Measure: Number; unit: Participants
Groups:
- Group II: Ustekinumab 45 mg: Partcipants received ustekinumab 45 mg at Weeks 0, 4 and 16. Treatments after Week 16 were dependent on clinical response. At Week 28, partcipants who achieved a greater than and equal 50 percentage but less than 75 percentage improvement in PASI were re-randomized to continue 45 mg every 12 week or dose adjust to 45 mg every 8 week dosing.
- Group III: Ustekinumab 90 mg: Partcipants received ustekinumab 90 mg at Weeks 0, 4 and 16. Treatments after Week 16 were dependent on clinical response. At Week 28, partcipants who achieved a greater than and equal 50 percentage but less than 75 percentage improvement in PASI were re-randomized to continue 90 mg every 12 week or dose adjust to 90 mg every 8 week dosing.
Arm/Group | Group I: Placebo | Group II: Ustekinumab 45 mg | Group III: Ustekinumab 90 mg
Number analyzed (Participants) | 410 | 409 | 411
Participants | 15 | 273 | 311
Statistical Analysis 1: Comparison: Group I: Placebo vs Group III: Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square; Stratified by baseline weight [less than or equal to 90 kg vs greater than 90 kg)]
Statistical Analysis 2: Comparison: Group I: Placebo vs Group II: Ustekinumab 45 mg; Null Hypothesis: No difference between ustekinumab 90 mg or 45 mg and placebo at an overall significance level of 0.05. Sample Size: With 1200 participants (400 in each treatment group), simulation studies were conducted to calculate the power to detect a treatment difference in the primary endpoint between ustekinumab groups and placebo using a CMH test stratified by baseline weight [<=90kg vs > 90 kg). For all the scenarios evaluated, the power is >99% at an overall significance level of 0.05; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square — To control for the multiplicity for the primary endpoint analysis, the Holm's procedure was used at an overall significance level of 0.05; Stratified by baseline weight [less than or equal 90 kg vs greater than 90 kg)]

2. Secondary Outcome: Number of Participants With Physician Global Assessment (PGA) of Cleared or Minimal at Week 12
Description: Number of participants achieving a physician global assessment (PGA) (0 [none] to 5 [severe]) of cleared or minimal at Week 12. The PGA is 7-point scale used in clinical trials of various diseases. In this the physician checks the state of the disease and gives them score from 0 (clear) to 5 (severe).
Time Frame: Week 12
Population: Intent to treat. All participants were included in the analysis according to the assigned treatment groups. Participant is considered a non- responder if the participant has used any pre-specified prohibited medications or discontinued due to lack of efficacy or had missing data at Week 12.
Measure: Number; unit: Participants
Groups:
- Group I: Placebo: Placebo partcipants received placebo at Weeks 0 and 4. At Weeks 12 and 16, placebo crossed over to receive ustekinumab 45 mg or 90 mg. Treatments after Week 16 were dependent on clinical response.
- Group III: Ustekinumab 90 mg: Partcipants received ustekinumab 90 mg at Weeks 0, 4 and 16. Treatments after Week 16 were dependent on clinical response. At Week 28, partcipants who achieved a greater than and equal to 50 percentage but less than 75 percentage improvement in PASI were re-randomized to continue 90 mg every 12 week or dose adjust to 90 mg every 8 week dosing.
Arm/Group | Group I: Placebo | Group II: Ustekinumab 45 mg | Group III: Ustekinumab 90 mg
Number analyzed (Participants) | 410 | 409 | 411
Participants | 18 | 277 | 300
Statistical Analysis 1: Comparison: Group I: Placebo vs Group III: Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square; Stratified by baseline weight [less than or equal 90 kg vs greater than 90 kg)]
Statistical Analysis 2: Comparison: Group I: Placebo vs Group II: Ustekinumab 45 mg; Null Hypothesis: No difference between ustekinumab 90 mg or 45 mg and placebo at an overall significancd level of 0.05; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel (CMH) chi square — To control the multiplicity for the primary and the secondary endpoint analyses, Holm's procedure was used but the two comparisons for the primary endpoint need to be significant first; Stratified by baseline weight [less than or equal 90 kg vs greater than 90 kg)]

3. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI) at Week 12
Description: Change in Dermatology Life Quality Index (DLQI) from baseline at Week 12. The DLQI is a 10-item questionnaire, that in addition to evaluating overall quality of life, can be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. Scores range from 0 (no impairment in quality of life) to 30 (most impairment in quality of life).
Time Frame: Baseline to Week 12
Population: Participants were included in the analysis according to the assigned treatment groups. Zero change is imputed if the partcipant has used any pre-specified prohibited medications or discontinued due to lack of efficacy. Other missing data were not imputed.
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Groups:
- Group II: Ustekinumab 45 mg: Participants received ustekinumab 45 mg at Weeks 0, 4 and 16. Treatments after Week 16 were dependent on clinical response. At Week 28, participants who achieved a greater than and equal 50 percentage but less than 75 percentage improvement in PASI were re-randomized to continue 45 mg every 12 week or dose adjust to 45 mg every 8 week dosing.
Arm/Group | Group I: Placebo | Group II: Ustekinumab 45 mg | Group III: Ustekinumab 90 mg
Number analyzed (Participants) | 400 | 401 | 402
Units on a scale | -0.5 [-4.0 to 3.0] | -8.0 [-14.0 to -4.0] | -9.0 [-14.0 to -5.0]
Statistical Analysis 1: Comparison: Group I: Placebo vs Group III: Ustekinumab 90 mg; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores; Analysis of variance on van der Waerden normal scores (Conover, 1980) with treatment and baseline weight (≤ 90kg vs > 90 kg) as factors in the model
Statistical Analysis 2: Comparison: Group I: Placebo vs Group II: Ustekinumab 45 mg; Null Hypothesis: No difference between ustekinumab 90 mg or 45 mg and placebo at an overall significance level of 0.05; Test type: Superiority or Other; p < 0.001, ANOVA on van der Waerden normal scores — To control the multiplicity for the primary and the secondary endpoint analyses, Holm's procedure was used but the two comparisons for the primary endpoint and the two comparisons for the 1st second endpoint analyses need to be significant first; Analysis of varianceon van der Waerden normal scores (Conover, 1980) with treatment and baseline weight (≤90 kg vs >90 kg) as factors in the model

4. Secondary Outcome: Number of Participants Visits With Psoriasis Area and Severity Index (PASI) 75 From Week 40 Through Week 52
Description: Number of visits at which participants randomized at Week 28 achieved at least 75 percent improvement from baseline in PASI from Week 40 through Week 52 in participants randomized at Week 28. PASI is a widely used tool for the measurement of severity of psoriasis. This is a test of how bad a person's psoriasis is. The scale combines redness, scaling, and thickness, as well as overall body involvement to determine the PASI score. The scale ranges from 0 (best) to 72 (worst).
Time Frame: Week 40 to Week 52
Population: All participants randomized at Week 28 were included in the analysis according to the assigned treatment groups. Participant is considered a non- responder if the participant has used any pre-specified prohibited medications or discontinued due to lack of efficacy.
Measure: Median (Inter-Quartile Range); unit: Participants
Groups:
- Group 1: Ustekinumab 45mg Every 8 Weeks: Participants received ustekinumab 45 mg at Weeks 0, 4, 16, 28, 36 and 44.
- Group 2: Ustekinumab 45mg Every 12 Weeks: Participants received ustekinumab 45 mg at Weeks 0, 4, 16, 28 and 40.
- Group 3: Ustekinumab 90 mg Every 8 Weeks: Participants received ustekinumab 90 mg at Weeks 0, 4, 16., 28, 36 and 44.
- Group 4: Ustekinumab 90 mg Every 12 Weeks: Participants received ustekinumab 90 mg at Weeks 0, 4, 16, 28 and 40.
- Group 5: Combined (8 Week Dosing): Combined Groups 1 and 3 (dosing every 8 weeks)
- Group 6: Combined (12 Week Dosing): Combined Groups 2 and 4 (dosing every 12 weeks)
Arm/Group | Group 1: Ustekinumab 45mg Every 8 Weeks | Group 2: Ustekinumab 45mg Every 12 Weeks | Group 3: Ustekinumab 90 mg Every 8 Weeks | Group 4: Ustekinumab 90 mg Every 12 Weeks | Group 5: Combined (8 Week Dosing) | Group 6: Combined (12 Week Dosing)
Number analyzed (Participants) | 45 | 48 | 32 | 33 | 77 | 81
Participants | 0 [0.0 to 2.0] | 1 [0.0 to 3.0] | 3 [1.5 to 4.0] | 1 [0.0 to 4.0] | 2 [0.0 to 4.0] | 1 [0.0 to 3.0]
Statistical Analysis 1: Comparison: Group 5: Combined (8 Week Dosing) vs Group 6: Combined (12 Week Dosing); Test type: Superiority or Other; p = 0.468, Cochran-Mantel-Haenszel (row mean score); Stratified by baseline weight [less than or equal to 90 kg vs greater than 90 kg)]
Statistical Analysis 2: Comparison: Group 1: Ustekinumab 45mg Every 8 Weeks vs Group 2: Ustekinumab 45mg Every 12 Weeks; Test type: Superiority or Other; p = 0.210, Cochran-Mantel-Haenszel (row mean score); Stratified by baseline weight [less than or equal to 90 kg vs greater than 90 kg)]
Statistical Analysis 3: Comparison: Group 3: Ustekinumab 90 mg Every 8 Weeks vs Group 4: Ustekinumab 90 mg Every 12 Weeks; Null Hypothesis: No difference between combined q8 group and the combined q12 group, 45 mg q8 and 45 mg q12, 90 mg q8 and 90 mg q12 at an overall significance level of 0.05; Test type: Superiority or Other; p = 0.014, Cochran-Mantel-Haenszel (row mean score) — To control the overall multiplicity, the combined groups was tested first and each dose will then be tested; but the primary and the 1st 2 secondary endpoint analyses need to be significant before this endpoint can be tested; Stratified by baseline weight [less than or equal to 90 kg vs greater than 90 kg)]

ADVERSE EVENTS:
Time Frame: Week 264
Description: 4 patients in the Ustekinumab 45 mg (after CP) and 7 patients in the Ustekinumab 90 mg (after CP) groups, discontinued study medication during the CP but had follow-up after CP and hence are included in the tables of frequent adverse events and serious adverse events after CP.
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP) | Placebo -> Ustekinumab 45 mg (After CP) | Placebo -> Ustekinumab 90 mg (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Serious Adverse Events (participants affected / at risk) | 8/410 | 8/409 | 5/411 | 40/197 | 41/195 | 81/407 | 73/409
Other Adverse Events (participants affected / at risk) | 116/410 | 119/409 | 114/411 | 168/197 | 159/195 | 342/407 | 343/409
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=410) | Ustekinumab 45 mg (CP) (N=409) | Ustekinumab 90 mg (CP) (N=411) | Placebo -> Ustekinumab 45 mg (After CP) (N=197) | Placebo -> Ustekinumab 90 mg (After CP) (N=195) | Ustekinumab 45 mg (After CP) (N=407) | Ustekinumab 90 mg (After CP) (N=409)
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 2
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 2 | 2 | 6 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 3 | 1 | 5 | 3
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Salivary gland calculus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 1 | 2 | 2 | 7
Cyst (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Device breakage (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hernia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cryptogenic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaphylactoid reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 2 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 3 | 1 | 1 | 2
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Genitourinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Open fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 1 | 2 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glomus tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 2 | 3
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Benign intracranial hypertension (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Complicated migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Substance abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 3 | 0 | 4 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 2
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ovarian torsion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pityriasis rubra pilaris (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alcohol detoxification (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Arterial stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Intra-abdominal haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=410) | Ustekinumab 45 mg (CP) (N=409) | Ustekinumab 90 mg (CP) (N=411) | Placebo -> Ustekinumab 45 mg (After CP) (N=197) | Placebo -> Ustekinumab 90 mg (After CP) (N=195) | Ustekinumab 45 mg (After CP) (N=407) | Ustekinumab 90 mg (After CP) (N=409)
Diarrhoea (Gastrointestinal disorders) | 11 | 9 | 11 | 13 | 7 | 35 | 27
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 2 | 10 | 6 | 17 | 13
Toothache (Gastrointestinal disorders) | 2 | 3 | 4 | 3 | 10 | 9 | 17
Injection site erythema (General disorders) | 1 | 6 | 6 | 5 | 5 | 17 | 23
Bronchitis (Infections and infestations) | 6 | 3 | 2 | 22 | 20 | 50 | 36
Gastroenteritis (Infections and infestations) | 2 | 4 | 2 | 13 | 13 | 43 | 35
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1 | 10 | 6 | 14 | 15
Influenza (Infections and infestations) | 2 | 3 | 4 | 25 | 19 | 42 | 48
Nasopharyngitis (Infections and infestations) | 29 | 30 | 28 | 69 | 75 | 137 | 143
Pharyngitis (Infections and infestations) | 3 | 1 | 5 | 7 | 9 | 18 | 21
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 10 | 6 | 5 | 12
Sinusitis (Infections and infestations) | 4 | 3 | 5 | 25 | 16 | 29 | 53
Upper respiratory tract infection (Infections and infestations) | 14 | 18 | 12 | 59 | 53 | 112 | 111
Urinary tract infection (Infections and infestations) | 3 | 0 | 3 | 7 | 7 | 15 | 23
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 8 | 8 | 21 | 18
Laceration (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 10 | 6 | 14 | 17
Muscle strain (Injury, poisoning and procedural complications) | 4 | 3 | 2 | 16 | 12 | 17 | 17
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 6 | 11 | 14 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 14 | 10 | 21 | 18 | 40 | 60
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 3 | 7 | 22 | 23 | 51 | 45
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1 | 9 | 5 | 22 | 29
Headache (Nervous system disorders) | 17 | 19 | 19 | 21 | 21 | 43 | 51
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 10 | 4 | 14 | 14
Depression (Psychiatric disorders) | 0 | 3 | 2 | 11 | 7 | 22 | 17
Insomnia (Psychiatric disorders) | 3 | 3 | 2 | 14 | 7 | 18 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 4 | 16 | 18 | 36 | 36
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 8 | 6 | 17 | 16 | 14
Hypertension (Vascular disorders) | 6 | 5 | 4 | 32 | 20 | 50 | 51

LIMITATIONS AND CAVEATS:
The count of patients with any nonserious adverse event (NAE) excludes patients who only had NAE that occured in <=5% of patients. This information may vary from existing approved labeling and publications due to the requirements of this website.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the PI is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.